CLINICAL TRIAL: NCT02073981
Title: Japan-First-in Large Scale Observational Study for Non-motor Symptoms and Treatment in Parkinson's Disease Patients.
Brief Title: Observational Study for Non-motor Symptoms and Treatment in Parkinson's Disease Patients
Acronym: J-FIRST
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: J-FIRST
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson Disease

SUMMARY:
This study is implemented to identify factors having an impact on improvement or exacerbation of non-motor symptoms, to provide information contributing to development of medical care in this field and improvement of patients' QOL, and to clarify the association between the use of istradefylline and non-motor symptoms or QOL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have wearing off under treatment with levodopa-containing drugs administered at least three times daily
* Patients who have at least one non-motor symptom as a complication
* Patients at least 20 years of age at the time of consent
* Patients who have given written consent
* Patients who are receiving outpatient care

Exclusion Criteria:

* Patients with dementia or a score of 23 or less on the Mini-Mental State Examination (MMSE)
* Patients, in the opinion of the investigator or subinvestigator, having conditions impairing the proper assessment of the MDS-UPDRS or PDQ-8 (e.g., patients who are receiving treatment for malignant tumor)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson Disease
Sampling Method: Non-Probability Sample
Enrollment: 1021 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Changing of Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 52 weeks
  MDS-UPDRS score will be collected from all registrant at each visit and on the last day of survey.
Changing of Parkinson's Disease Questionaire-8 (PDQ-8) score. | 52 weeks
  PDQ-8 score will be collected from all registrant at each visit and on the last day of survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Juntendo University Hospital, Bunkyo-ku, Tokyo, Japan